CLINICAL TRIAL: NCT05112536
Title: A Phase 2, Open-Label, Single-Arm Study of Single-Dose Lead-In and Neoadjuvant Trilaciclib and Chemotherapy in Patients With Early-Stage Triple Negative Breast Cancer (TNBC)
Brief Title: Trilaciclib, a CDK4/6 Inhibitor, in Patients With Early-Stage Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G1T28-212
Record Dates: First submitted 2021-10-06; First posted 2021-11-09 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-12

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer
Keywords: Breast Cancer; Triple Negative Breast Cancer; CDK4/6 Inhibitor; trilaciclib dihydrochloride; Cosela; Immuno-oncology; Solid tumor; Chemotherapy-induced myelosuppression; Myeloprotective; Cyclin-dependent kinase 4/6 inhibitor; Neoadjuvant; HER2-negative; TNBC; Breast cancer surgery; Trilaciclib; Myeloprotection; pembrolizumab; carboplatin; doxorubicin; cyclophosphamide; Dose-dense anthracycline/cyclophosphamide; paclitaxel; Chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — trilaciclib; Cyclophosphamide; Doxorubicin; Paclitaxel; Carboplatin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trilaciclib plus chemotherapy (Experimental): Trilaciclib lead-in, followed by trilaciclib plus anthracycline/cyclophosphamide, then trilaciclib plus taxane chemotherapy:
  * Lead-in trilaciclib (240mg/m2) single dose monotherapy
  * Trilaciclib (240mg/m2) + doxorubicin (60 mg/m2) + cyclophosphamide (600 mg/m2) + pembrolizumab (per Investigator discretion; 400mg)
  * Trilaciclib (240mg/m2) + paclitaxel (80 mg/m2) + carboplatin (per Investigator discretion; AUC 1.5)
  Interventions: Drug: Trilaciclib; Drug: Cylophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Carboplatin (Investigator discretion); Biological: Pembrolizumab (Investigator discretion)

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib is administered IV as monotherapy during the lead-in phase and administered prior to chemotherapy on each day chemotherapy is administered during the treatment phase.
  Other Names: COSELA®; G1T28
Drug: Cylophosphamide — Cyclophosphamide administered IV every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Other Names: CYTOXAN®
Drug: Doxorubicin — Doxorubicin administered as an IV bolus every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Other Names: ADRIAMYCIN®
Drug: Paclitaxel — Paclitaxel administered weekly for the last 12 cycles (cycles 5-16), each cycle 1 week in length.
  Other Names: TAXOL®
Drug: Carboplatin (Investigator discretion) — Carboplatin, if given, is administered IV weekly at the start of paclitaxel administration, for the last 12 cycles (cycles 5-16).
  Other Names: PARAPLATIN®
Biological: Pembrolizumab (Investigator discretion) — Pembrolizumab, if given, is administered IV every 6 weeks throughout the treatment phase (cycles 1, 4, 9, 15).
  Other Names: KEYTRUDA®

SUMMARY:
The purpose of this study is to evaluate the mechanism of action, as well as the safety and efficacy of trilaciclib in combination with standard of care treatment in the neoadjuvant setting of early-stage triple negative breast cancer (TNBC).

This study will have four phases: 1) Screening Phase, 2) Trilaciclib Lead-In Phase, 3) Treatment Phase, and 4) Surgery and Follow-Up Phase. After a screening phase of up to 21 day, each participant will receive trilaciclib single-dose monotherapy during the lead-in phase, followed by a tumor biopsy. During the treatment phase, each participant will receive trilaciclib with standard of care chemotherapy. Immunotherapy may be included during the treatment phase, per standard of care. 3-5 weeks following conclusion of the treatment phase, each participant will undergo definitive surgery. A 30-day Safety Follow-up Visit will occur 30 days after the last dose of trilaciclib and an End of Study Visit will occur within 14 days after definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Suitability of therapy and patient intends to undergo curative surgery
* Documented diagnosis of estrogen receptor (ER)-negative and progesterone receptor (PR)-negative tumor
* Primary tumor ≥ 1.5 cm with any nodal status
* Provide archival tissue for the baseline tissue sample
* ECOG performance status of 0 or 1
* Demonstrates adequate organ function
* Research tumor biopsies including at least one on-treatment biopsy (and additional biopsy at baseline, if required)
* Participants of child bearing potential must be willing to use 2 forms of contraception during the study and for 6 months following study treatment

Exclusion Criteria:

* Prior systemic therapies or radiation for current breast cancer
* History of invasive malignancy ≤3 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* History of breast cancer including ipsilateral ductal carcinoma in situ (DCIS) treated with radiotherapy at any time
* Previous exposure to doxorubicin of more than 200 mg/m2 (as lifetime exposure to doxorubicin is not to exceed 450 mg/m2)
* For patients who will receive pembrolizumab:

  * History of active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy is not considered a form of systemic treatment
  * Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drugs
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Known history of active tuberculosis (Bacillus Tuberculosis)
* History of severe hepatic impairment
* Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure (Class II-IV as defined by the New York Heart Association [NYHA] functional classification system)
* Known history of stroke, cerebrovascular accident, severe/unstable angina, myocardial infarction, or coronary angioplasty/stenting/bypass grafting within 6 months prior to enrollment
* Known serious active infection (e.g., human immunodeficiency virus [HIV], hepatitis B or C, tuberculosis).
* Women who are pregnant or breastfeeding
* Participation in other studies involving active treatment with investigational drug(s)
* Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA Department of Medicine - Hematology/Oncology, Santa Monica, California
  - PIH Health, Whittier, California
  - Nebraska Hematology-Oncology, P.C., Lincoln, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 7 clinical locations, including academic, community, and hospital network locations. Recruitment occurred between November 2021 and August 2022. The first participant was enrolled on March 3rd, 2022. The last participant was enrolled on August 2nd, 2022.
Pre-assignment Details: 24 participants were enrolled. As an open-label study, all participants received trilaciclib during the monotherapy, lead-in phase, followed by trilaciclib plus doxorubicin/cyclophosphamide and paclitaxel (AC/T). Additions of pembrolizumab and/or carboplatin were at physician discretion.
Groups:
- Trilaciclib Plus Chemotherapy: All subjects received trilaciclib lead-in (240mg/m2) single dose monotherapy, followed by trilaciclib plus anthracycline/cyclophosphamide (Trilaciclib (240mg/m2) + doxorubicin (60 mg/m2) + cyclophosphamide (600 mg/m2) + pembrolizumab (per Investigator discretion; 400mg)), then trilaciclib plus taxane chemotherapy (Trilaciclib (240mg/m2) + paclitaxel (80 mg/m2) + carboplatin (per Investigator discretion; AUC 1.5) + pembrolizumab (per Investigator discretion; 400mg).
  Trilaciclib: Trilaciclib is administered IV as monotherapy during the lead-in phase and administered prior to chemotherapy on each day chemotherapy is administered during the treatment phase.
  Cylophosphamide: Cyclophosphamide administered IV every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Doxorubicin: Doxorubicin administered as an IV bolus every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Paclitaxel: Paclitaxel administered weekly for the last 12 cycles (cycles 5-16), each cycle 1 week in length.
  Carboplatin (Investigator discretion): Carboplatin, if given, is administered IV weekly at the start of paclitaxel administration, for the last 12 cycles (cycles 5-16).
  Pembrolizumab (Investigator discretion): Pembrolizumab, if given, is administered IV every 6 weeks throughout the treatment phase (cycles 1, 4, 9, 15).
Period: Overall Study
Arm/Group | Trilaciclib Plus Chemotherapy
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trilaciclib Plus Chemotherapy
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 57.0 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.88 (9.219)
Stage at diagnosis [Count of Participants; unit: Participants] — For Stage I - Stage III, cancer is present. The higher the number, the bigger the tumor size and the more it has spread into nearby tissues.
  * Stage I - cancer is present but is limited to the place where it started; also referred to as early-stage cancer.
  * Stage II - cancer is present and has spread to nearby tissue
  * Stage III - cancer is present and has spread to nearby tissue with a larger tumor than Stage II
  Participants
    Stage I | 2
    Stage II | 19
    Stage III | 3
Histologic Grade [Count of Participants; unit: Participants] — Per the American Cancer society, cancer cells are given a grade when removed from the breast and checked in a lab. Grading is determined by how much the cancer cells look like normal cells. Grading is used to predict outcome (prognosis) and to help the doctor determine the best course of treatment.
  * Grade I - cancer is slower-growing and less likely to spread
  * Grade 2 - cancer is grower faster than Grade 1 but slower than Grade 3
  * Grade 3 - faster-growing cancer that's more likely to spread
  Participants
    Grade 1 | 1
    Grade 2 | 3
    Grade 3 | 20
Histopathological type at diagnosis [Count of Participants; unit: Participants] — Histopathological typing is completed by looking at the morphology, or the size, shape, location, and structure, of cancer cells under a microscope. A biopsy, or a procedure to remove tissue or cells for testing, is undergone to obtain cells to view. Cancer tissue with lobular carcinomas generally have cells in a single-file line and occur in fatty tissue, where ductal carcinomas have cells which re-form glandular structures and are generally more likely to create a mass.
  Participants
    Ductal | 20
    Lobular | 1
    Other | 3
BRCA Mutation Status [Count of Participants; unit: Participants]
  Negative | 10
  BRCA 1 | 1
  BRCA 2 | 0
  BRCA 1/2 | 1
  Not done/Other | 12
PD-L1 status [Count of Participants; unit: Participants]
  Positive | 1
  Negative | 2
  Not done/Unknown | 21
Easter Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants] — ECOG Performance Scale measures how cancer impacts a patient's daily activities. A higher score indicates a lower ability to function independently and the patient's cancer is having a significant impact on their day-to-day activities. For this trial, scores of 0 to 1 were required to participate, indicating a patient was fully active or able to carry out work of a light or sedentary nature. The scale goes from 0 (fully active) to 5 (deceased).
  Participants
    0 | 22
    1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Immune-based Mechanism of Action
Description: Evaluated 7 days after a single-dose of trilaciclib, measured by the change in CD8+ T cells/regulatory T cells (Treg) ratio in tumor tissue; post-trilaciclib ratio minus pre-trilaciclib ratio.
  Research shows a correlation between immune cells, (tumor-infiltrating lymphocytes - TILs), and favorable outcomes. Both the presence of effector CD8+ T cells and the ratio of effector CD8+ T cells to immune-suppressive regulatory T cells (Treg) correlate with improved outcome and long-term survival in solid cancers. Therefore, the higher the ratio of CD8+ T cells/Tregs, the better the predicted outcome for a patient. This outcome measure is completed by looking at tumor tissue under a microscope.
Time Frame: Up to 8 days after lead-in trilaciclib dose
Population: Full Analysis Set 1 (FAS1), defined as all enrolled participants who received trilaciclib during the Trilaciclib Lead-in Phase, for whom pre-trilaciclib and post-trilaciclib monotherapy biopsies were available for analysis.
Measure: Median (Inter-Quartile Range); unit: CD8+/Tregs ratio
Groups:
- Trilaciclib Plus Chemotherapy: Trilaciclib lead-in, followed by trilaciclib plus anthracycline/cyclophosphamide, then trilaciclib plus taxane chemotherapy:
  * Lead-in trilaciclib (240mg/m2) single dose monotherapy
  * Trilaciclib (240mg/m2) + doxorubicin (60 mg/m2) + cyclophosphamide (600 mg/m2) + pembrolizumab (per Investigator discretion; 400mg)
  * Trilaciclib (240mg/m2) + paclitaxel (80 mg/m2) + carboplatin (per Investigator discretion; AUC 1.5) + pembrolizumab (per Investigator discretion; 400mg)
  Trilaciclib: Trilaciclib is administered IV as monotherapy during the lead-in phase and administered prior to chemotherapy on each day chemotherapy is administered during the treatment phase.
  Cylophosphamide: Cyclophosphamide administered IV every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Doxorubicin: Doxorubicin administered as an IV bolus every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Paclitaxel: Paclitaxel administered weekly for the last 12 cycles (cycles 5-16), each cycle 1 week in length.
  Carboplatin (Investigator discretion): Carboplatin, if given, is administered IV weekly at the start of paclitaxel administration, for the last 12 cycles (cycles 5-16).
  Pembrolizumab (Investigator discretion): Pembrolizumab, if given, is administered IV every 6 weeks throughout the treatment phase (cycles 1, 4, 9, 15).
Arm/Group | Trilaciclib Plus Chemotherapy
Number analyzed (Participants) | 23
CD8+/Tregs ratio | 0.3 [-0.5 to 2.7]
Statistical Analysis 1: Comparison: Trilaciclib Plus Chemotherapy; Test type: Other; p = 0.101, Wilcoxon signed-rank test

2. Secondary Outcome: Pathologic Complete Response (pCR) Rate
Description: Rate of pCR using the definition of ypT0/Tis ypN0 (i.e., no invasive residual tumor in breast or nodes; noninvasive breast residuals allowed) as assessed by the local pathologist.
Time Frame: Up to 26 weeks
Population: Full Analysis Set (FAS), enrolled participants who received at least one dose of any study drug during the treatment period, where treatment period consists of Trilaciclib Lead-in Phase and the Treatment Phase.
Measure: Count of Participants; unit: Participants
Groups:
- Trilaciclib Plus Chemotherapy: Trilaciclib lead-in, followed by trilaciclib plus anthracycline/cyclophosphamide, then trilaciclib plus taxane chemotherapy:
  * Lead-in trilaciclib (240mg/m2) single dose monotherapy
  * Trilaciclib (240mg/m2) + doxorubicin (60 mg/m2) + cyclophosphamide (600 mg/m2) + pembrolizumab (per Investigator discretion; 400mg)
  * Trilaciclib (240mg/m2) + paclitaxel (80 mg/m2) + carboplatin (per Investigator discretion; AUC 1.5)+ pembrolizumab (per Investigator discretion; 400mg)
  Trilaciclib: Trilaciclib is administered IV as monotherapy during the lead-in phase and administered prior to chemotherapy on each day chemotherapy is administered during the treatment phase.
  Cylophosphamide: Cyclophosphamide administered IV every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Doxorubicin: Doxorubicin administered as an IV bolus every 2 weeks for the first 4 cycles (1-4), each cycle 2 weeks in length.
  Paclitaxel: Paclitaxel administered weekly for the last 12 cycles (cycles 5-16), each cycle 1 week in length.
  Carboplatin (Investigator discretion): Carboplatin, if given, is administered IV weekly at the start of paclitaxel administration, for the last 12 cycles (cycles 5-16).
  Pembrolizumab (Investigator discretion): Pembrolizumab, if given, is administered IV every 6 weeks throughout the treatment phase (cycles 1, 4, 9, 15).
Arm/Group | Trilaciclib Plus Chemotherapy
Number analyzed (Participants) | 24
Participants
  Achieved pCR | 10
  Did not achieve pCR | 14

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Safety/tolerability as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: Up to 28 weeks
Population: Full Analysis Set 2 (FAS2), included enrolled patients who had received at least one dose of a study drug during the Treatment Phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib Plus Chemotherapy
Number analyzed (Participants) | 24
Participants
  Adverse Events CTCAE grade >/= 3 | 15
  Adverse Events CTCAE grade >/= 4 | 5
  Study drug related adverse event | 24
  Study drug related serious adverse event | 2
  Trilaciclib-related adverse event leading to discontinuation | 0
  Adverse event leading to death | 0
  Trilaciclib adverse events of special interest (AESI) | 10

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: The statistical analysis plan pre-specified the collection of adverse events for all participants as a single arm/group irrespective of intervention
Groups:
- Trilaciclib Plus Chemotherapy: All subjects received trilaciclib lead-in (240mg/m2) single dose monotherapy, followed by trilaciclib plus anthracycline/cyclophosphamide (Trilaciclib (240mg/m2) + doxorubicin (60 mg/m2) + cyclophosphamide (600 mg/m2) + pembrolizumab (per Investigator discretion; 400mg)), then trilaciclib plus taxane chemotherapy (Trilaciclib (240mg/m2) + paclitaxel (80 mg/m2) + carboplatin (per Investigator discretion; AUC 1.5) + pembrolizumab (per Investigator discretion; 400mg).
  This trial investigated the mechanism of action of trilaciclib, and not safety profile comparison between trilaciclib treated patients receiving or not receiving pembrolizumab, nor comparison of the safety profile between trilaciclib treated subjects receiving or not receiving carboplatin. This was a single-arm study; only 1 treatment arm/group was prospectively defined. Therefore safety was reported in accordance to the study design (i.e., a single arm/group). Additionally, 21 of 24 subjects enrolled were treated with pembrolizumab and 21 of 24 patients enrolled were treated with carboplatin. Thus, the safety reporting as a single group is representative of the vast majority of participants (21/24 (87.5%)).
Arm/Group | Trilaciclib Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib Plus Chemotherapy (N=24)
Abscess limb (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Herpes simplex encephalitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Physical deconditioning (General disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib Plus Chemotherapy (N=24)
Nausea (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Vomitting (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 21
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 4
Catheter site pain (General disorders) | 3
Oedema (General disorders) | 3
Pain (General disorders) | 3
Auxillary pain (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Catheter site erythema (General disorders) | 1
Catheter site pruritis (General disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Injection site pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Thirst (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 17
Pruritis (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 5
Nail discolouration (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Onychclasis (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2
Restless leg syndrome (Nervous system disorders) | 2
Ageusia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Ophthalmic migraine (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Oral herpes (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Eye infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increase (Investigations) | 2
White blood cell count decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Protein total decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 6
Adjustment disorder (Psychiatric disorders) | 1
Irritabiliy (Psychiatric disorders) | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hot flush (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 2
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Embolism (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Lacrimation increased (Eye disorders) | 3
Vision blurred (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Cataract (Eye disorders) | 1
Eye ulcer (Eye disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Vulvovaginal dryness (Reproductive system and breast disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Glycosuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
A limitation of this study was the small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to submit any disclosure to Sponsor for review at least thirty (30) days prior to submission. Within sixty (60) days of its receipt, Sponsor can provide feedback on any disclosure Sponsor may require Investigator to remove, Confidential Information (other than study data), and/or to delay the proposed publication or presentation for an additional sixty (60) days to enable Sponsor to seek patent protection for inventions.

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT05112536/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT05112536/SAP_001.pdf